CLINICAL TRIAL: NCT02083133
Title: Dosing Strategies in Diabetic Patients With End Stage Renal Disease (ESRD) or Hemodialysis (DOSE-HD Study)
Brief Title: Insulin Dosing in Diabetic Patients With End Stage Renal Disease (ESRD) or Hemodialysis
Acronym: DOSE-HD
Status: Completed | Type: Observational
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Pete Antonopoulos, Clinical Pharmacist- Principal Investigator, Cook County Health
Other Study IDs: 13-188
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Diabetes; Hypoglycemia; Renal Dysfunction; Insulin Dosing
Keywords: Diabetes; Renal Failure; Dialysis; End Stage Renal Disease; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Renal Insufficiency; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- End Stage Renal Disease: GFR 15 ml/min or less or on Dialysis
- Chronic Kidney Disease Stage 4: GFR 15-30 ml/min
- Chronic Kidney Disease Stage -3: GFR 30-60 ml/min

SUMMARY:
The purpose of this study is to assess whether the current recommendation for a 50% dose reduction in insulin for diabetic patients with a creatinine clearance (CrCl) ≤15 mL/min or on hemodialysis results in an increased number of hypoglycemic episodes.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient men and women 18 years of age and older with a diagnosis of type 2 diabetes mellitus (T2DM) with CrCl ≥60, 16-59 or ≤15 milliliters/minute.

Exclusion Criteria:

* Patients less than 18 years of age, pregnant patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In patient hospitalized greater than or equal to three days, diabetic with CKD 3-5 or on dialysis on insulin therapy
Sampling Method: Probability Sample
Enrollment: 496 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia | Last 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pete Antonopoulos, PharmD, Principal Investigator — Cook County Hospital
Locations (1):
- John H Stroger Hospital of Cook County, Chicago, Illinois, United States